CLINICAL TRIAL: NCT02050516
Title: Randomized Controlled Comparison of Single Embryo Culture Versus Group Culture Using a Micro-well Group Culture Dish in Humans
Brief Title: Comparison of Single vs Group Embryo Culture in Micro-well Group Culture Dish
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elif Güler Ergin (Other)
Collaborators: Vitrolife (Industry)
Responsible Party: Sponsor-Investigator, Elif Güler Ergin, MD, Eurofertil IVF Health Center
Organization: Eurofertil IVF Health Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: WOW-1
Record Dates: First submitted 2014-01-29; First posted 2014-01-30 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Infertility
Keywords: Blastocyst, micro-well group culture dish
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- single embryo culture (Active Comparator): single embryo culture in single drops inside micro-well group culture dish
  Interventions: Other: micro-well group culture dish
- group embryo culture (Experimental): group embryo culture in a single drop inside micro-well group culture dish
  Interventions: Other: micro-well group culture dish

INTERVENTIONS:
Other: micro-well group culture dish — an embryo culture dish containing nine micro-wells in the middle.

SUMMARY:
Does group culture using micro-well group culture dishes improve human blastocyst development compared to single embryo culture?

ELIGIBILITY:
Inclusion Criteria: female age uner 40, male age under 60 patients undergoing IVF-treatment with oocyte collection after ovarian hyperstimulation having signed the study-specific consent form patient fulfilling clinic's standard criteria for blastocyst culture minimum 5 normally fertilized oocytes at the time of fertilization check

Exclusion Criteria: use of any type of surgically retrieved sperm cells patients undergoing any kind of genetic diagnosis at any developmental stage

-

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Blastocyst development | 6 days

SECONDARY OUTCOMES:
Implantation rate | 1 month

OTHER OUTCOMES:
Clinical pregnancy rate | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Elif Güler Ergin, MD, Principal Investigator — Eurofertil IVF Health Center
Locations (1):
- Eurofertil IVF Health Center, Istanbul, Turkey (Türkiye)